CLINICAL TRIAL: NCT06097247
Title: Family Functioning and Adverse Side Effects of Family-based Therapy for Anorexia Nervosa. User Perspectives and Observed Changes - a Mixed Method Explorative Study Designed to Inform a Clinical Trial Testing Treatment Improvements
Brief Title: Family Functioning and Adverse Side Effects of Family-based Therapy for Anorexia Nervosa
Acronym: Spor3
Status: Active, not recruiting | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Foreningen Spiseforstyrrelser og Selvskade (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-21041874
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Anorexia in Adolescence; Anorexia in Children; Family Relations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study examines potential adverse side effects on family functioning and parent-child relationships of standard treatment family-based therapy (FBT) for anorexia nervosa (AN) in children and youths.

DETAILED DESCRIPTION:
Background:

Family-based treatment (FBT) for anorexia nervosa (AN) in children and youth has contributed significantly to the treatment of a disorder that has otherwise had a poor prognosis. Focus in FBT is on empowering parents to take full control over their child's nourishment. However, many parents are concerned how FBT might affect the relationship with their child as parents assume a double role of insisting on eating and weight gain, while at the same time providing emotional support, when this distresses the child. Moreover, FBT may have a "blind eye" to psychological difficulties with e.g. emotion regulation and interpersonal challenges, and thus inadvertently exacerbating them while focusing narrowly on eating and weight gain.

Aim:

The aim of the study is to quantitatively investigate side-effects of FBT by:

1. Assessing average changes as well as variations across families from start of FBT, after 3 months, and at end of FBT in four domains: perceived parental stress level and family function, emotion regulation ability and perceived attachment to parents.
2. Qualitatively describe the lived experience of young persons as well as parents going through FBT.
3. Based on the results of a) and b) to generate hypotheses on which additions and / or alterations to treatment that may mitigate potential adverse side effects of FBT- treatment. These modifications to FBT will be tested in a future clinical trial.

Exploratively, we will investigate whether level of family functioning at three months of FBT predicts changes in the four above mentioned domains at end of treatment (EOT), thus identify early in treatment the families at risk of adverse side-effects of FBT.

Methods:

Family functioning, parental stress level and attachment perception are measured with questionnaires only. Emotion regulation is measured with questionnaires and the Tangram Puzzle Task. The qualitative section of the study consists of interviews at end of treatment and will be conducted in a co-operation with the Danish patient organization Eating Disorders and Self Harm.

The project is a sub study to the larger study investigating response to treatment of eating disorders in youth: Effectiveness of Family-based Intervention in a Child and Adolescent Mental Health Service (CAMHS) for Children and Adolescents With Eating Disorders (VIBUS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of F50.0 or F50.1 first time of treatment with family-based treatment living with a minimum of one parent informed consent from young person and parents

Exclusion Criteria:

* non Danish-speaking

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All eligible patients presenting for treatment in the region are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The Systemic Clinical Outcome and Routine Evaluation - 15 items version (SCORE-15). | Start and End of Treatment (an average of 1 year).
  Minimum value: 1 Maximum value: 5 Higher scores mean worser outcome.
The Kerns Security Scale-Revised 21 | Start and End of Treatment (an average of 1 year).
  Minimum value: 1 Maximum value: 4 Higher scores indicate more secure attachment.
Difficulties in Emotion Regulation Scale (DERS) | Start and End of Treatment (an average of 1 year).
  Minimum value: 1 Maximum value: 5 Higher scores mean worser outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Katrine Pagsberg, professor, Principal Investigator — Child and Adolescent Mental Health Care Centre, Capital Region of Denmark
Locations (1):
- Child and Adolescent Mental Health Care Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No